CLINICAL TRIAL: NCT06956703
Title: NAZA - Nottingham/Astra ZenecA Prospective IBD Cohort Study
Acronym: NAZA
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22GA031
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-12

CONDITIONS: Gastro-Intestinal Disorder; Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Digestive System Diseases; Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Crohn's Disease - anti-TNFα therapy: Consultant will prescribe biologic dose, frequency and duration as normal standard of care
- Crohn's Disease - ustekinumab: Consultant will prescribe biologic dose, frequency and duration as normal standard of care
- Crohn's Disease - upadacitinib: Consultant will prescribe biologic dose, frequency and duration as normal standard of care
- Ulcerative Colitis - anti-TNFα therapy: Consultant will prescribe biologic dose, frequency and duration as normal standard of care
- Ulcerative Colitis - vedolizumab: Consultant will prescribe biologic dose, frequency and duration as normal standard of care
- Control non-IBD: No biologic will be prescribed

SUMMARY:
The goal of this observational study is to learn about the comparisons of inflammatory markers between IBD and non-IBD (control) participants.

The main question it aims to answer is:

Are there differences in inflammatory markers between IBD and non-IBD (control) participants.

DETAILED DESCRIPTION:
A cohort study in patients with moderate to severely active Crohns Disease (CD) and Ulcerative Colitis (UC) who are switching to new targeted biologic therapy (with a different mode of action) - onto either anti-TNFα therapy or vedolizumab for UC or onto anti-TNFα therapy or ustekinumab or upadacitinib for CD and undergoing routine endoscopic assessments as part of normal clinical practice.

The investigator will also recruit participants without these conditions (controls) who are due for a lower GI colonoscopy as part of the UK national bowel cancer screening programme or on any hospital/ medical/ clinical screening list or any other appropriate list with no pathology found on examination.

CD & UC patients will provide blood and stool samples at 3 timepoints (baseline, 3mths, 12mths) as well as extra tissue biopsies taken at standard care endoscopies within 12mths. Controls will provide a blood sample and stool sample as well as extra tissue biopsies taken at standard care colonoscopies.

Samples will be analysed to characterise any observable traits (phenotype) and molecular variability in patients which may be associated with clinical response to the treatment.

The investigator hopes the information gained from this study may help improve the understanding of Inflammatory Bowel Diseases (IBD) and help to develop better ways of treating the condition and predicting the course of the disease and how patients may respond to different treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent before any study specific procedures

AND

2a. Patients of at least 16 years of age with active Crohn's disease defined as: CRP > = 5 mg/L OR FCP > = 250 μg/g OR Visible ulcerations on ileocolonoscopy with a total SES-CD > = 7, or > = 4 if disease is confined to the terminal ileum OR visable active disease on cross-sectional imaging. Are switching to a new mechanism of action (MOA) onto anti-TNF therapy or ustekinumab or upadacitinib

OR

2b. Patients of at least 16 years (no upper age limit) with active UC defined as: CRP > = 5 mg/L OR FCP > = 250 μg/g OR Mayo endoscopy subscore > = 2. Are switching to a new mechanism of action (MOA) onto either anti-TNFα therapy or vedolizumab

OR

2c. Non-IBD participants who are attending for a lower GI colonoscopy at any participating site. On any hospital/ medical/ clinical screening list or any other appropriate list with no pathology found on examination.

Exclusion Criteria:

1. Inability to give informed consent
2. Any positive result from previous screening for serum hepatitis B surface antigen, hepatitis C or human immunodeficiency virus (HIV)
3. An ongoing infection requiring treatment
4. Clinical evidence of active COVID infection and/or evidence of active COVID determined by local standard care procedures
5. Participation in a clinical study with pharmacological intervention within 3 months prior to Baseline visit.
6. Current diagnosis of cancer
7. Having received a solid organ or stem cell transplant
8. Having received a transfusion of blood, plasma, or platelets within 120 days prior to enrolment
9. Confirmed pregnancy at time of enrolment
10. For non-IBD participants: A prior history of IBD (CD, UC, microscopic colitis, indeterminate colitis or IBD unspecified)
11. Clinical judgement by the investigator that the patient should not participate in the study
12. Under 16yrs of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A cohort study in patients with moderate to severely active Crohn's Disease (CD) and Ulcerative Colitis (UC) who are switching to new targeted biologic therapy (with a different mode of action) - onto either anti-TNFα therapy or vedolizumab for UC or onto anti-TNFα therapy or ustekinumab or upadacitinib for CD and undergoing routine endoscopic assessments as part of normal clinical practice.
  We will also recruit participants without these conditions (controls) who are due for a lower GI colonoscopy as part of the UK national bowel cancer screening programme or on any hospital/ medical/ clinical screening list or any other appropriate list with no pathology found on examination.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The comparison of the IL-23/Th17 inflammatory axis between IBD and healthy control samples | Baseline, Month 3 and Month 12

SECONDARY OUTCOMES:
Characterisation of IL-23/Th17 inflammatory axis within IBD biosamples stratified by prior biologic exposure | Baseline, Month 3 and Month 12
Comparison of mRNA sequencing readouts, characterisation of tissue and immune cell populations, characterisation of protein expression and characterisation of microbial species in the stool and tissue | Baseline, Month 3 and Month 12
  The above will be stratified by disease type and status, demographic features of the participant, biologic exposure, clinical and endoscopic response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Moran Professor, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom